CLINICAL TRIAL: NCT05506046
Title: Messages About Reduced Nicotine in Combusted Tobacco Products: An Online Randomized Controlled Trial
Brief Title: Messages About Reduced Nicotine in Combusted Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Lyudmila Popova, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H22639
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Health Communication; Smoking; Smoking, Tobacco; Smoking Behaviors; Risk Behavior
MeSH Terms: conditions — Smoking; Tobacco Smoking; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reduced Nicotine Messages (Experimental): Participants will receive messages with information about reduced nicotine cigarettes.
  Interventions: Behavioral: Reduced nicotine message exposure
- Modified Risk Messages (Experimental): Participants will receive messages with information about e-cigarettes.
  Interventions: Behavioral: Modified risk message exposure
- Combined Message -- Reduced Nicotine + Modified Risk Exposure (Experimental): Participants will receive messages about reduced nicotine cigarettes and about e-cigarettes.
  Interventions: Behavioral: Combined message exposure (reduced nicotine + modified risk)
- Control (Other): Participants will receive messages about bottled water which should have no impact on the outcomes of interest.
  Interventions: Behavioral: Control message exposure

INTERVENTIONS:
Behavioral: Reduced nicotine message exposure — Participants will be shown two messages about harms of reduced nicotine cigarettes. The two messages will be drawn from a pool of five messages. The messages will communicate that reduced nicotine cigarettes will still have the rest of the harmful chemicals and cause diseases as the regular cigarettes, but they would make it easier to quit.
  Arms: Reduced Nicotine Messages
Behavioral: Modified risk message exposure — Participants will be shown two messages about electronic cigarettes as an alternative to regular cigarettes. The two messages will be drawn from a pool of five messages. The messages will communicate that electronic cigarettes are less likely than regular cigarettes to cause severe diseases such as lung cancer.
  Arms: Modified Risk Messages
Behavioral: Combined message exposure (reduced nicotine + modified risk) — Participants will be shown two messages, one from the reduced nicotine message set and one modified risk message set.
  Arms: Combined Message -- Reduced Nicotine + Modified Risk Exposure
Behavioral: Control message exposure — Participants will be shown two messages about drinking bottled water. These will be selected from a pool of five message. The messages display specific water products and describe hydration as a healthy activity.
  Arms: Control

SUMMARY:
The investigators will conduct a message-exposure experiment with nationally representative samples of smokers, dual-users (cigarettes and e-cigarettes), and young adult non-smokers (aged 18-29).

Experimental messages will address the reduction of nicotine in cigarettes. Participants will also complete a follow-up survey after 2 weeks, measuring their recall of the messages and behaviors since message exposure.

DETAILED DESCRIPTION:
A national probability-based sample will be recruited to include 900 current exclusive smokers, 450 dual users, and 450 young adult (18-29) non-smokers, evenly split between men and women.

The study will be conducted using a self-administered, online questionnaire via proprietary, web-assisted interviewing software.

Participants are randomized to one of four conditions:

* reduced nicotine messages
* modified risk messages
* a combination of reduced nicotine message and modified risk message
* control messages with no cigarette-related content

Participants will take part in two sessions: in session 1 (estimated at about 15 min) participants will see the messages and report immediate outcomes including risk perceptions.

In session 2, which will take place 2 weeks after session 1, participants will complete a brief 5-minute survey measuring their recall of the messages and behaviors since message exposure.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older:
* Belonging to one of three groups of participants; 900 current exclusive smokers, 450 dual users (cigarettes and e-cigarettes), and 450 young adult (18-29) non-smokers, evenly split between men and women.
* Enrolled in existing nationally representative panel where recruitment is based

Exclusion Criteria:

- None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1901 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pei D, Reynolds RM, Ntansah CA, Hackworth EE, Henderson KC, Yang B, Duong HT, Ashley DL, Thrasher JF, Popova L. Independent and combined effects of very low nicotine cigarette messages and e-cigarette messages: a randomised clinical trial. Tob Control. 2025 Dec 19;34(e1):e48-e56. doi: 10.1136/tc-2023-058556. PMID 38664002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a panel. Participants were pre-identified based on internal data on age and smoking status: adults who exclusively smoked cigarettes, adults who dual used cigarettes and e-cigarettes, and young adults (aged 18-29) who never smoked.
Pre-assignment Details: The panel sample (probability sample) included 971 adults who smoked exclusively, 240 adults who dual used cigarettes and e-cigarettes, and 458 young adults (18-29 years old) who never smoked. To augment the sample of adults who dual used, additional participants were recruited from the opt-in, non-probability sample (n=232) bringing the total sample size to 1901.
Period: Overall Study
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Started (Number of participants who started session 1) | 468 | 484 | 476 | 473
Compete Session 1 (Number of participants who completed session 1) | 468 | 484 | 476 | 473
Started Session 2 (Number of participants who started session 2) | 379 | 383 | 374 | 374
Completed (number of participants who completed session 2) | 379 | 383 | 374 | 374
Not Completed | 89 | 101 | 102 | 99
Not completed — Lost to Follow-up | 89 | 101 | 102 | 99

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control | Total
Number analyzed (Participants) | 468 | 484 | 476 | 473 | 1901
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 128 | 141 | 134 | 147 | 550
  30-44 years | 105 | 110 | 114 | 112 | 441
  45-59 years | 119 | 112 | 106 | 108 | 445
  60+ | 116 | 121 | 122 | 106 | 465
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 262 | 259 | 240 | 1016
  Male | 213 | 222 | 217 | 233 | 885
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 328 | 314 | 348 | 321 | 1311
  Black, non-Hispanic | 49 | 63 | 52 | 61 | 225
  Other, non-Hispanic | 20 | 19 | 11 | 21 | 71
  Hispanic | 55 | 63 | 46 | 54 | 218
  Two Races or more, non-Hispanic | 16 | 25 | 19 | 16 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 468 | 484 | 476 | 473 | 1901

OUTCOME MEASURES:

1. Primary Outcome: Perceived Health Risk of VLNCs (Absolute)
Description: Measured with a single item, assesses participant's perception of own risk of overall harm to health under conditions of smoking reduced nicotine cigarettes every day. Response options range from 1 (Not at all likely) to 5 (Extremely likely), with higher scores representing a better outcome. An additional option, "Don't know", is also provided.
Time Frame: Immediately after exposure
Population: The number of participants analyzed included all participants in each condition who responded to the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 418 | 427 | 420 | 428
score on a scale | 4.09 [3.99 to 4.19] | 3.81 [3.71 to 3.90] | 4.03 [3.93 to 4.13] | 3.87 [3.78 to 3.97]

2. Secondary Outcome: Interest in Trying Reduced Nicotine Cigarettes
Description: A single item measuring how interested a participant is in trying reduced nicotine cigarettes. Response options are from 1 (not at all) to 7 (extremely), with higher scores representing a worse outcome. An additional option, "Don't know", is also provided.
Time Frame: Immediately after exposure
Population: The number of participants analyzed included all participants in each condition who responded to the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 432 | 442 | 449 | 440
score on a scale | 3.09 [2.89 to 3.28] | 2.95 [2.76 to 3.14] | 3.08 [2.90 to 3.27] | 3.15 [2.95 to 3.34]

3. Secondary Outcome: Intention to Switch From Cigarettes to Electronic Nicotine Products
Description: A single item measuring intention (during the next 6 months) to switch completely from cigarettes to electronic nicotine products. Response options are from 1 (not at all likely) to 7 (extremely likely), with higher scores representing a better outcome. An additional option, "Don't know", is also provided.
Time Frame: Immediately after exposure
Population: The number of participants analyzed included participants who 1) are adults who smoked exclusively and adults who dual used and 2) responded to the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 324 | 340 | 335 | 332
score on a scale | 3.15 [2.96 to 3.33] | 2.97 [2.79 to 3.15] | 2.91 [2.73 to 3.09] | 2.86 [2.68 to 3.05]

4. Secondary Outcome: Perceived Addictiveness of VLNCs
Description: A single item measuring participants' perception of likelihood of developing addiction to reduced nicotine cigarettes under conditions of smoking them every day. Response options are from 1 (Not at all likely) to 5 (Extremely likely), with higher scores representing a worse outcome. An additional option, "Don't know", is also provided.
Time Frame: Immediately after exposure
Population: The number of participants analyzed included all participants in each condition who responded to the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 404 | 416 | 411 | 406
score on a scale | 3.68 [3.58 to 3.78] | 3.74 [3.64 to 3.84] | 3.65 [3.55 to 3.75] | 3.71 [3.61 to 3.82]

5. Secondary Outcome: VLNC Comparative Risk Perceptions
Description: A single item measuring perceptions of comparative risk of smoking reduced nicotine cigarettes vs regular cigarettes. Response options are from 1 (Much less harmful) to 5 (Much more harmful), with higher scores representing a better outcome. An additional option, "Don't know", is also provided.
Time Frame: Immediately after exposure
Population: The number of participants analyzed included all participants in each condition who responded to the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 393 | 401 | 413 | 404
score on a scale | 2.97 [2.90 to 3.04] | 2.81 [2.74 to 2.88] | 2.89 [2.82 to 2.96] | 2.78 [2.71 to 2.85]

6. Secondary Outcome: VLNC Policy Support
Description: A single item measuring support for the policy to reduce nicotine by 95% in all cigarettes. Response options are from 1 (Strongly Oppose) to 5 (Strongly Support), with higher scores representing a better outcome. An additional option, "Don't know", is also provided.
Time Frame: Immediately after exposure
Population: The number of participants analyzed included all participants in each condition who responded to the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 447 | 447 | 446 | 450
score on a scale | 3.20 [3.09 to 3.32] | 3.08 [2.96 to 3.19] | 3.21 [3.09 to 3.32] | 3.14 [3.03 to 3.26]

7. Secondary Outcome: Perceived Message Effectiveness
Description: A three-item scale measuring to what extent participants think the messages they saw discourage them from wanting to smoke, make smoking seem unpleasant, and make them concerned about health risks of smoking.
  Response options: from 1 (Disagree) to 4 (Neither Disagree nor Agree) to 7 (Strongly Agree).
  Higher scores represent a better outcome. The final perceived message effectiveness score is the mean of the response to the three items.
Time Frame: Immediately after exposure
Population: The number of participants analyzed included all participants who responded to all three outcome measures.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 468 | 484 | 476 | 471
score on a scale | 4.55 [4.41 to 4.70] | 3.98 [3.84 to 4.13] | 4.32 [4.17 to 4.46] | 2.33 [2.18 to 2.47]

8. Secondary Outcome: Perceived Health Risk of VLNCs (Absolute) at Post-test
Description: as for outcome 1
Time Frame: Two weeks after exposure
Population: The analysis population included participants in each condition that responded to the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 300 | 300 | 304 | 300
score on a scale | 3.68 [3.57 to 3.80] | 3.62 [3.51 to 3.74] | 3.68 [3.56 to 3.79] | 3.62 [3.50 to 3.73]

9. Secondary Outcome: Smoking Behavior
Description: Single item measuring the average number of cigarettes smoked per day in the past two weeks.
Time Frame: Two weeks after exposure
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: number of cigarettes/day
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
Number analyzed (Participants) | 287 | 284 | 284 | 281
number of cigarettes/day | 11.64 [10.60 to 12.68] | 11.97 [10.93 to 13.02] | 12.78 [11.74 to 13.83] | 11.97 [10.92 to 13.02]

ADVERSE EVENTS:
Time Frame: Low risk study, no adverse events data collected.
Description: Low risk study, no adverse events data collected.
Arm/Group | Reduced Nicotine Messages | Modified Risk Messages | Combined Message -- Reduced Nicotine + Modified Risk Exposure | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT05506046/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT05506046/ICF_001.pdf